CLINICAL TRIAL: NCT02147015
Title: Personalized Variable Versus Fixed Dose Corticosteroids Therapy in Hospitalized Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Personalized Variable Versus Fixed Dose Glucocorticoid Therapy in AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Guoqiang Cao,MD, Vice Chair of Department of Respiratory Medicine, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIP
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute Exacerbations; Corticosteroids; Chronic Obstructive Pulmonary Disease; Doses
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glucocorticoids; Methylprednisolone; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized variable dose of glucocorticoids arm (Experimental): Use of personalized variable dose of glucocorticoids according to a rating scale starting from the first day of hospitalization for 5 days, together with other necessary treatments, including antibiotics, Inhaled corticosteroid (ICS), long-acting beta2-agonist (LABA), Long-Acting Muscarinic Antagonists(LAMA), short-acting beta2-agonist (SABA), and other physical treatments.
  Interventions: Drug: Glucocorticoids; Drug: Antibiotics; Drug: Inhaled corticosteroid (ICS); Drug: Long-Acting Muscarinic Antagonists(LAMA); Drug: Short-acting beta2-agonist (SABA); Other: Physical treatments; Drug: long-acting beta2-agonist (LABA)
- Fixed dose of glucocorticoids arm (Other): Use of fixed term of glucocorticoids (40mg) starting from the first day of hospitalization for 5 days, together with other necessary treatments, including antibiotics, ICS, LABA, LAMA, SABA, and other physical treatments.
  Interventions: Drug: Glucocorticoids; Drug: Antibiotics; Drug: Inhaled corticosteroid (ICS); Drug: Long-Acting Muscarinic Antagonists(LAMA); Drug: Short-acting beta2-agonist (SABA); Other: Physical treatments; Drug: long-acting beta2-agonist (LABA)

INTERVENTIONS:
Drug: Glucocorticoids
  Other Names: methylprednisolone
Drug: Antibiotics
Drug: Inhaled corticosteroid (ICS)
Drug: Long-Acting Muscarinic Antagonists(LAMA)
Drug: Short-acting beta2-agonist (SABA)
Other: Physical treatments
Drug: long-acting beta2-agonist (LABA)

SUMMARY:
The hypothesis is that in acute exacerbated Chronic Obstructive Pulmonary Disease (AECOPD), personalized variable dose glucocorticoid treatment will result in superior clinical outcome when compared to fixed dose therapy.

DETAILED DESCRIPTION:
Treatment with glucocorticoid for acute exacerbations of COPD results in the improvement of clinical outcomes. However, the optimal doses of glucocorticoid for each individual patient has not been determined. According to GOLD Report 2014, a dose of 40 mg prednisone per day for 5 days is recommended (Evidence B), although there are insufficient data to provide firm conclusions concerning the optimal duration of corticosteroid therapy of acute exacerbations of COPD. The purpose of the current study is to compare clinical outcomes of personalized or fixed dose of glucocorticoid in patients with acute exacerbations of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation of COPD as defined by the presence of at least 2 of the following: change in baseline dyspnea, cough, or sputum quantity or purulence.

Exclusion Criteria:

* Signs of severe exacerbation (arterial pH < 7.26 or PaCO2 > 9.3 kPa)
* History of asthma
* Significant or unstable co-morbidity
* Participated in another study 4 weeks before admission
* Previously randomized to this study
* Known hypersensitivity to prednisolone
* Inability to give written informed consent
* Radiological diagnosis of pneumonia
* Estimated survival of less than 6 months due to severe comorbidity
* Use of glucocorticoid within 1 month before admission

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 6 months
  1. death from any cause;
  2. admission to the intensive care unit;
  3. readmission to the hospital because of COPD
  4. the necessity to intensify pharmacologic treatment during in-hospital (due to persistence of dyspnoea, bronchospasm, or worsening of other respiratory symptoms)

SECONDARY OUTCOMES:
length of hospital stay | 1 month

OTHER OUTCOMES:
Hospital costs | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Guoqiang Cao, Medical Doctor, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Davies L, Angus RM, Calverley PM. Oral corticosteroids in patients admitted to hospital with exacerbations of chronic obstructive pulmonary disease: a prospective randomised controlled trial. Lancet. 1999 Aug 7;354(9177):456-60. doi: 10.1016/s0140-6736(98)11326-0. PMID 10465169
- [Background] Lindenauer PK, Pekow PS, Lahti MC, Lee Y, Benjamin EM, Rothberg MB. Association of corticosteroid dose and route of administration with risk of treatment failure in acute exacerbation of chronic obstructive pulmonary disease. JAMA. 2010 Jun 16;303(23):2359-67. doi: 10.1001/jama.2010.796. PMID 20551406
- [Background] Leuppi JD, Schuetz P, Bingisser R, Bodmer M, Briel M, Drescher T, Duerring U, Henzen C, Leibbrandt Y, Maier S, Miedinger D, Muller B, Scherr A, Schindler C, Stoeckli R, Viatte S, von Garnier C, Tamm M, Rutishauser J. Short-term vs conventional glucocorticoid therapy in acute exacerbations of chronic obstructive pulmonary disease: the REDUCE randomized clinical trial. JAMA. 2013 Jun 5;309(21):2223-31. doi: 10.1001/jama.2013.5023. PMID 23695200
- [Derived] Li L, Zhao N, Ma X, Sun F, He B, Qin Z, Wu K, Wang X, Zhao Q, Zhang S, Nie N, Luo D, Sun B, Shen Y, He Y, Wen F, Zheng J, Jones P, Cao G. Personalized Variable vs Fixed-Dose Systemic Corticosteroid Therapy in Hospitalized Patients With Acute Exacerbations of COPD: A Prospective, Multicenter, Randomized, Open-Label Clinical Trial. Chest. 2021 Nov;160(5):1660-1669. doi: 10.1016/j.chest.2021.05.024. Epub 2021 May 21. PMID 34023318